# **Protocol Synopsis – Public Summary Version**

For: NCT06381986

A Clinical Study on the Safety and Efficacy of SHJ002 Sterile Ophthalmic Solution in the Treatment of Corneal Erosion in Patients with Sjogren's Syndrome

Sponsor: Sunhawk Vision Biotech, Inc.

IRB Approval Date: December 16, 2024

Document Date: December 16, 2024 (Final IRB-approved version: Protocol v2.0, dated

October 30, 2024)

## 1. Study Objectives

Primary Objective:

To evaluate the efficacy of SHJ002 ophthalmic solution in reducing corneal fluorescein staining in patients with corneal erosion secondary to Sjogren's Syndrome.

Secondary Objectives:

To assess changes in regional fluorescein staining (iCFS) and patient-reported symptoms using the SANDE questionnaire.

### 2. Study Design

Design: Multicenter, double-blinded, randomized, vehicle-controlled, parallel-group Phase 2

trial

Participants: Adults ≥18 years with Sjogren's Syndrome and corneal erosion

Randomization: 1:1 ratio to SHJ002 or vehicle group Treatment: One drop per eye, twice daily for 12 weeks

Sites: Multiple hospitals in Taiwan

## 3. Endpoints

**Primary Endpoint:** 

Change from Baseline to Week 12 in Total Corneal Fluorescein Staining (NEI Scale, score range 0–15; higher scores indicate more severe staining)

Secondary Endpoints:

- Change in Inferior Corneal Fluorescein Staining (iCFS) Score by NEI Scale (0–3 per region; higher scores = worse outcome)
- Change in Symptom Assessment in Dry Eye (SANDE) score (0-100 scale; higher = worse symptoms)

#### 4. Inclusion / Exclusion Criteria

#### **Key Inclusion:**

- Adults ≥18 years
- Diagnosed with Sjogren's Syndrome and corneal erosion
- Negative pregnancy test for women of childbearing potential

#### **Key Exclusion:**

- Ocular diseases other than corneal erosion/DED
- Recent ocular surgery
- Conflicting medication use or other interfering conditions

# **5. Statistical Analysis Overview**

Primary Efficacy Analysis:

Mixed Model for Repeated Measures (MMRM) used to analyze change in CFS from baseline, with covariates including treatment, visit, interaction, and baseline score.

Reporting:

Least squares means (LSM), standard error (SE), 95% confidence intervals (CI), and treatment group comparisons with p-values.

Missing Data:

Assumed Missing at Random (MAR); no imputation was needed.

This is a summary protocol document prepared specifically for public registration purposes on ClinicalTrials.gov. Proprietary scientific or commercial details have been redacted.